CLINICAL TRIAL: NCT00655512
Title: Comparison of Skin Thickness Under Treatment With Pimecrolimus 1% Cream (Elidel® 1% Cream), Hydrocortisonacetat 1% Cream (Hydrogalen® Cream), Betamethasonvalerat 0,1% Cream (Betagalen® Cream) and Clobetasol-17-propionat 0,05% Cream (Clobegalen® Cream) Assessed by Optical Coherence Tomography (OCT) and 20-MHZ Ultrasound - a Single Blind, Placebo-controlled, Randomized, Monocenter Clinical Trial
Brief Title: Comparison of Skin Thickness Under Treatment With Pimecrolimus 1% Cream, Hydrocortisonacetat 1% Cream, Betamethasonvalerat 0,1% Cream and Clobetasol-17-propionat 0,05% Cream Assessed by Optical Coherence Tomography (OCT) and 20-MHZ Ultrasound
Acronym: OCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TUD-OCT011-023
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: pimecrolimus; hydrocortison; betamethasone; clobetasol-17-Propionat; Optical Coherence Tomography; skin healthy probands
MeSH Terms: interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Active Comparator)
  Interventions: Drug: hydrocortisonacetat 1% cream; Drug: betamethasonvalerat 0,1% cream; Drug: clobetasol-17-propionat 0,05% cream
- 2 (Active Comparator)
  Interventions: Drug: pimecrolimus 1% cream; Drug: betamethasonvalerat 0,1% cream; Drug: clobetasol-17-propionat 0,05% cream
- 3 (Active Comparator)
  Interventions: Drug: pimecrolimus 1% cream; Drug: hydrocortisonacetat 1% cream; Drug: clobetasol-17-propionat 0,05% cream
- 4 (Active Comparator)
  Interventions: Drug: pimecrolimus 1% cream; Drug: hydrocortisonacetat 1% cream; Drug: betamethasonvalerat 0,1% cream
- 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pimecrolimus 1% cream — twice a day one fingertip at the testareas (forehead and forearm/back of the hand) for 4 weeks
  Other Names: Elidel 1% cream
  Arms: 2; 3; 4
Drug: hydrocortisonacetat 1% cream — twice a day one fingertip at the testareas (forehead and forearm/back of the hand) for 4 weeks
  Other Names: Hydrogalen cream
  Arms: 1; 3; 4
Drug: betamethasonvalerat 0,1% cream — twice a day one fingertip at the testareas (forearm/back of the hand) for 4 weeks
  Other Names: Betagalen cream
  Arms: 1; 2; 4
Drug: clobetasol-17-propionat 0,05% cream — twice a day one fingertip at the testareas (forearm/back of the hand) for 4 weeks
  Other Names: Clobegalen cream
  Arms: 1; 2; 3
Drug: Placebo — twice a day one fingertip at the testareas (forehead and forearm/back of the hand) for 4 weeks
  Arms: 5

SUMMARY:
to compare the atrophogenic potentials of pimecrolimus 1% cream, hydrocortisonacetat 1% cream, betamethasonvalerat 0,1% cream and clobetasol-17-Propionat 0,05% cream

ELIGIBILITY:
Inclusion Criteria:

* male and female probands age between 18-40 years
* skin healthy
* skintype I-III according to Fitzpatrick

Exclusion Criteria:

* women of childbearing potential without adequate contraception
* pregnant or breastfeeding
* genetic defect of epidermal barrier
* external or systemic treatment with drugs, which probably have an effect to the thickness of skin or to the production of teleangiektasien within the last 6 month before study entry
* skin disease, which hinder the evaluation with OCT, ultrasound or dermaphot
* UV treatment within the last 4 weeks before study entry
* participation to another clinical trial within the last 30 days before study entry
* allergy against pimecrolimus or hydrocortison or betamethasonvalerat or Clobetasol-17-propionat
* severe systemic diseases; ongoing immunosuppressive treatment
* planned vaccination should realize before study entry or 28 days after end of treatment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
thickness of epidermis | 9 times in 4 weeks

SECONDARY OUTCOMES:
atrophogenic effect assessed by dermaphot | 9 times in 4 weeks
moisture of skin assessed by corneometer | 9 times in 4 weeks
transpire of skin assessed by tewameter | 9 times in 4 weeks
thickness of dermis | 9 times in 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roland Aschoff, MD, Principal Investigator — Department of Dermatology, Medical Faculty, Technical University Dresden, Germany
Locations (1):
- Department of Dermatology, Medical Faculty, TU Dresden, Dresden, Germany